CLINICAL TRIAL: NCT01180621
Title: PCIRN Evaluation of Seasonal Trivalent Influenza Vaccine for 2010-2011 in Young Children in the First Year After the H1N1 Pandemic
Brief Title: Evaluation of Seasonal Influenza Vaccine for 2010-2011 in Young Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: IWK Health Centre (Other); Canadian Institutes of Health Research (CIHR) (Other Government); GlaxoSmithKline (Industry)
Responsible Party: Dr. Joanne Langley, Canadian Center for Vaccinology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PCIRN RT-07
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Seasonal Influenza
Keywords: vaccine; Seasonal Influenza Vaccine; Influenza Vaccine; Vaccine Safety; Vaccine Immunogenicity; Fluviral 2010-2011
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Eggs

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fluviral (Experimental): 0.25 mL Fluviral for children up to and including 35 months of age 0.50 mL Fluviral for children 36-59 months of age
  Interventions: Biological: Fluviral

INTERVENTIONS:
Biological: Fluviral — 0.25 mL Fluviral for children up to and including 35 months of age 0.50 mL Fluviral for children 36-59 months of age
  Other Names: Influenza Virus Vaccine; Trivalent, Inactivated; Split Virion; Prepared in Eggs

SUMMARY:
The seasonal influenza vaccination program for 2010-2011 will be the first to follow the H1N1 pandemic of 2009. Many children either had the H1N1 infection or the adjuvanted H1N1 vaccine. Both H1N1 infection and adjuvanted vaccine produced strong immune responses which could last for some time.

The seasonal influenza vaccine for this fall will be a trivalent inactivated product (regular seasonal influenza vaccine)once again, without adjuvant. It will contain 3 strains of killed, split-apart viruses that might circulate this winter, including the H1N1 pandemic strain. It is theoretically possible that giving the H1N1-containing seasonal vaccine to people who still have some immunity to H1N1 virus could result in more frequent side-effects. However, there is no good evidence that pre-existing immunity to a strain in the vaccine does increase side-effects. In short, there could be nothing out of the ordinary this fall but it would be prudent to check this before public flu vaccination programs begin.

DETAILED DESCRIPTION:
This study will assess the safety of seasonal influenza vaccination in children who received one or two doses of the adjuvanted H1N1 vaccine last year. It will also measure residual immunity to the H1N1 virus and immune responses to the seasonal vaccine. It will be carried out before the new vaccine is released for general use so that we have an accurate picture of vaccine safety and responses for other Canadians.

A total of 200 children (50 at each site) 12-59 month olds, are being asked to participate in this study. A research nurse will conduct a telephone screening with potential participants to determine if they are eligible for the study. Volunteers must have had one or two doses of the adjuvanted H1N1 vaccine before January 31, 2010. To eligible participants do not need a previous years seasonal flu vaccine(TIV)however, this will be recorded.

The study involves 1-2 vaccination visits 28 days apart. Those children who have not received a previous dose of TIV will receive a second dose at visit # 2. After each vaccination, there will be contacts 1 and 7 days later for a description of any symptoms experienced. A blood sample will be requested at at each study visit (2 or 3 visits depending on previous TIV history) to measure immune responses to the seasonal vaccine.

The study will take 21-42 days to complete, depending upon whether or not the child received a previous dose of seasonal TIV vaccination. The 4 study sites are in Vancouver, Calgary, Montreal and Halifax.

Each subject's parent will be asked to keep daily notes of any changes at the injection site (pain, redness, swelling) and any general symptoms (such as irritability, drowsiness, decreased appetite, sleep disturbance,sweating and shivering, including your axilla or rectal temperature, for 7 days after each vaccination. Major health changes will be assessed for 21 days post vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided for the subject by a parent or legal guardian.
* Subjects whose parents the investigator believes can and will comply with the requirements of the protocol (i.e. return for follow-up visits, record safety observations, able to converse with study personnel including by telephone).
* Age 12-59 months at Visit 1, male or female
* Receipt of one or two doses of Arepanrix (adjuvanted H1N12009 vaccine, GlaxoSmithKline (GSK)) in 2009 documented by written record or attested by a confident personal recollection (window for vaccination will be 1 October 2009 to January 31, 2010).

Exclusion Criteria:

* Systemic hypersensitivity to hens' eggs or to any other Fluviral S/F vaccine component such as thimerosal
* History of a life-threatening reaction to any influenza vaccine
* Receipt of Arepanrix after January 31st , 2010
* Receipt of non-study TIV (Trivalent Influenza Vaccine)for the 2010-2011 season
* Receipt of any live vaccine within 4 weeks or inactivated vaccine within one week of study entry or planned administration of any non-study vaccines during the study period
* Thrombocytopenia or any bleeding disorder that contraindicates IM injection or blood collection
* Receipt of blood or any blood-derived products within the past 3 months
* Chronic illness at a stage that could interfere with trial participation (stable health conditions are acceptable, such as diabetes, lung disease, heart conditions etc)
* Immune compromise as a result of a medical condition, transplantation or immunosuppressive medication, not including topical or aerosol medications
* Participation in any other research study involving a non-approved drug or medical device

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of 2010-2011 seasonal trivalent influenza vaccine (TIV) | 7 days
  Assessing reactogenicity on days 1-6 following TIV administration.

SECONDARY OUTCOMES:
To measure immune response to each component of TIV. | 42 days
  Determining if there is a relationship between pre-TIV influenza haemagglutinin titers (ie, 6 to 10 months after receipt of adjuvanted vaccine), post TIV titers, and reactogenicity following TIV receipt.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Langley, MD, Principal Investigator — Dalhousie University
Locations (4):
- Canada (4):
  - ACHIEVE Research, Alberta Children's Hospital, Calgary, Alberta
  - Vaccine Evaluation Center, Vancouver, British Columbia
  - Candian Center for Vaccinology, Dalhousie University, Halifax, Nova Scotia
  - McGill University Health Centre - Vaccine Study Centre, Montreal, Quebec

REFERENCES:
- [Derived] Langley JM, Scheifele DW, Quach C, Vanderkooi OG, Ward B, McNeil S, Dobson S, Kellner JD, Kuhn S, Kollman T, MacKinnon-Cameron D, Smith B, Li Y, Halperin SA. Safety and immunogenicity of 2010-2011 H1N12009-containing trivalent inactivated influenza vaccine in children 12-59 months of age previously given AS03-adjuvanted H1N12009 pandemic vaccine: a PHAC/CIHR Influenza Research Network (PCIRN) study. Vaccine. 2012 May 14;30(23):3389-94. doi: 10.1016/j.vaccine.2012.03.046. Epub 2012 Mar 30. PMID 22469860